CLINICAL TRIAL: NCT00002571
Title: Study of Promace-Cytabom With Trimethoprim Sulfamethoxazole, Zidovudine (AZT), and Granulocyte Colony Stimulating Factor (G-CSF) in Patients With AIDS-Related Lymphoma, Phase II
Brief Title: SWOG-9320 Combination Chemotherapy, Radiation Therapy, and Antiviral Therapy in Treating Patients With AIDS-Related Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000063620; SWOG-9320 (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 1999-11-01; First posted 2004-05-24 (Estimated); Last update posted 2013-01-24 (Estimated); Status verified 2013-01

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma; AIDS-related diffuse mixed cell lymphoma; AIDS-related diffuse small cleaved cell lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Bleomycin; Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Cytarabine; Doxorubicin; Etoposide; Leucovorin; Methotrexate; Prednisone; Trimethoprim, Sulfamethoxazole Drug Combination; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ProMACE-CytaBOM + G-CSF (Experimental): 6 cycles of 21 days each of ProMACE-CytaBOM (cyclophosphamide 490 mg/m^2 on day 1, doxorubicin 19 mg/m^2 on day 1, etoposide 90 mg/m^2 on day 1, cytarabine 225 mg/m^2 on day 8, bleomycin 5 u/m^2 on day 8, methotrexate 90 mg/m^2 on day 8, leucovorin 25 mg/m^2 q 6 hours on days 8-9, vincristine 1.4 mg/m^2 on day 8, prednisone 60 mg/m^2 on days 1-14, allopurinol 300 mg on days 1-21 of cycle 1 and days 1-8 of cycle 2 only) plus 1 double strength tablet TMP/SMX 3 days a week plus G-CSF 5 ug/kg on days 9-20. Patients also receive intrathecal cytarabine 30 mg/m^2 (BM positive: 5 doses spaced evenly during 1st 2 cycles, then on day 1 of cycles 3-6; CSF cytology positive: 5 doses spaced evenly during 1st cycle, then on day 1 of cycles 2-6; BM and CSF negative: 5 doses spaced evenly within 1 month of completion of cycle 6). All patients with CR or PR after systemic therapy and IT cytarabine receive 2400 cGy RT to the whole brain in 12 fractions.
  Interventions: Biological: bleomycin sulfate; Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: doxorubicin hydrochloride; Drug: etoposide; Drug: leucovorin calcium; Drug: methotrexate; Drug: prednisone; Drug: trimethoprim-sulfamethoxazole; Drug: vincristine sulfate; Radiation: radiation therapy; Drug: Intrathecal cytarabine

INTERVENTIONS:
Biological: bleomycin sulfate — 5u/m2 IV Q21days x 6 cycles
Biological: filgrastim — 5ug/kg SC, Days 9-20, Q 21 days x 6 cycles
  Other Names: G-CSF
Drug: cyclophosphamide — 490 mg/m2 IV Q 21 days x 6 cycles
Drug: cytarabine — 225 mg/m2 IV Q 21 days x 6 cycles
Drug: doxorubicin hydrochloride — 19 mg/m2 IV Q 21 days x 6 cycles
Drug: etoposide — 90 mg/m2 IV Q 21 days x 6 cycles
  Other Names: VP-16
Drug: leucovorin calcium — 25 mg/m2 po 24 hours after methotrexate Q 6 hours x 4 doses for 6 cycles.
Drug: methotrexate — 90 mg/m2 IV, Q 21 days x 6 cycles.
Drug: prednisone — 60 mg/m2 po QD x 14days for 6 cycles
Drug: trimethoprim-sulfamethoxazole — 1 double throughout strength treatment tablet po on Monday, Wednesday, and Friday x 6, 21 day cycles
  Other Names: TMP/SMX
Drug: vincristine sulfate — 1.4 mg/m2 IV Q 21 Days x 6 cycles
Radiation: radiation therapy — All patients achieving a CR or PR following systemic therapy and IT Ara-C, will receive 2,400 cGy in two hundred cGy fractions to the whole brain. Fields should adequately encompass all meningeal surfaces.
Drug: Intrathecal cytarabine — If initial bone marrow positive:
  Ara-C 30 mg/m2 IT per dose x 5 doses spaced evenly during the first two cycles of therapy. Ara-C 30 mg/m2 IT Day 1 of each subsequent cycle.
  If initial CSF cytology positive:
  Ara-C 30 mg/m2 IT per dose x 5 doses spaced evenly during the first cycle of therapy. If CSF negative after above, Ara-C 30 mg/m2 IT Day 1 of each subsequent cycle. If CSF positive after initial five doses of Ara-C, IT MTX 12 mg per dose x 5 doses should be given spaced evenly during the second cycle of therapy.
  If initial bone marrow and CSF negative:
  Ara-C 30 mg/m2 IT per dose x 5 doses to be given spaced evenly within 1 month of completion of systemic therapy.
  Other Names: IT Ara-C

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Antiviral therapy may be effective treatment for AIDS-related lymphoma.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy, radiation therapy, and antiviral therapy in treating patients who have AIDS-related lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Assess the response rate of AIDS-related lymphoma to ProMACE-CytaBOM (cyclophosphamide, doxorubicin, etoposide, prednisone, cytarabine, bleomycin, vincristine, methotrexate). II. Assess the toxic effects of ProMACE-CytaBOM in patients with AIDS-related lymphoma. III. Evaluate whether the incorporation of filgrastim (G-CSF) into the regimen allows treatment with full doses of the myelotoxic agents in these patients. IV. Determine whether intensive CNS treatment with intrathecal cytarabine and whole-brain irradiation prevents meningeal relapse or controls meningeal lymphomatous involvement in these patients.

OUTLINE: Patients are stratified according to participating institution and descriptive factors: histopathology (diffuse large cleaved/noncleaved and immunoblastic lymphomas vs all others), CD4 count (less than 50 vs 50 or more cells/mm3), prior opportunistic infection (yes vs no), performance status (0 and 1 vs 2), concurrent AZT (yes vs no), concurrent protease inhibitors (yes vs no), marrow involvement (yes vs no). Patients receive ProMACE-CytaBOM regimen as follows: Cyclophosphamide, doxorubicin, and etoposide IV on day 1 Cytarabine, bleomycin, vincristine, and methotrexate IV on day 8 Oral prednisone on days 1-14 Oral leucovorin calcium every 6 hours for 4 doses on day 9 Patients also receive filgrastim (G-CSF) subcutaneously on days 9-20 and oral co-trimoxazole 3 days a week throughout treatment, plus antiretroviral therapy at the discretion of the treating physician. Treatment repeats every 21 days for a maximum of 6 courses. Patients with progressive disease are removed from study after 2 courses. Remaining patients receive an additional 2 treatment courses and are then restaged. Patients without stable or progressive disease receive 2 more courses in the absence of unacceptable toxicity. Patients with positive bone marrow at study entry receive CNS prophylaxis with 5 evenly spaced doses of intrathecal cytarabine during the first 2 treatment courses and on day 1 of each subsequent course. Patients with positive CSF cytology at study entry receive intrathecal cytarabine on days 1-5 of the first treatment course and on day 1 of each subsequent course if CSF negative after 5 daily doses. Patients whose CSF remains positive after 5 days receive 5 evenly spaced doses of intrathecal methotrexate during the second treatment course. Patients with negative bone marrow and CSF cytology at study entry receive 5 evenly spaced doses of intrathecal cytarabine within 1 month of systemic therapy. All patients achieving a complete or partial response following systemic therapy and intrathecal cytarabine receive cranial irradiation to all meningeal surfaces. Patients are followed monthly for 1 year, every 2 months for 1 year, every 3 months for 1 year, then annually thereafter.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study over approximately 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically proven intermediate or high grade non-Hodgkin's lymphoma of one of the following histologies: Follicular, predominantly large cell Diffuse, small cleaved cell Diffuse mixed, small and large cell Diffuse, large cell (cleaved or noncleaved) Immunoblastic, large cell Small noncleaved cell, Burkitt's or non-Burkitt's No lymphoblastic lymphoma Prior diagnosis of AIDS or HIV positivity required Confirmation of HIV antibody status by Western blot mandatory Bidimensionally measurable or evaluable disease No primary CNS lymphoma Concurrent registration on protocol SWOG-8947 (central serum repository) required

PATIENT CHARACTERISTICS: Age: Over 18 Performance status: SWOG 0-2 Hematopoietic: Absolute neutrophil count at least 500/mm3 Platelet count at least 75,000/mm3 Hepatic: AST no greater than 1.5 times normal Alkaline phosphatase no greater than 1.5 times normal LDH no greater than 1.5 times normal PT/PTT normal Renal: Creatinine no greater than 2.0 times normal Creatinine clearance at least 60 mL/min Cardiovascular: No serious abnormalities on EKG No history of severe coronary artery disease No history of cardiomyopathy, congestive heart failure, or arrhythmia Other: No active uncontrolled infection No active second malignancy within 5 years except adequately treated nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix Not pregnant or nursing Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY: No prior chemotherapy or radiotherapy for lymphoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 1994-06; Primary Completion 2003-11 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Response | every 3 months while on protocol treatment

CONTACTS AND LOCATIONS:
Overall Officials: Lode J. Swinnen, MD, Study Chair — Loyola University
Locations (85):
- United States (85):
  - MBCCOP - University of South Alabama, Mobile, Alabama
  - CCOP - Greater Phoenix, Phoenix, Arizona
  - Veterans Affairs Medical Center - Phoenix (Hayden), Phoenix, Arizona
  - Veterans Affairs Medical Center - Tucson, Tucson, Arizona
  - Arizona Cancer Center, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Veterans Affairs Medical Center - Little Rock (McClellan), Little Rock, Arkansas
  - Veterans Affairs Medical Center - Long Beach, Long Beach, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Beckman Research Institute, City of Hope, Los Angeles, California
  - Veterans Affairs Outpatient Clinic - Martinez, Martinez, California
  - CCOP - Bay Area Tumor Institute, Oakland, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of California Davis Medical Center, Sacramento, California
  - CCOP - Santa Rosa Memorial Hospital, Santa Rosa, California
  - David Grant Medical Center, Travis Air Force Base, California
  - Veterans Affairs Medical Center - Denver, Denver, Colorado
  - University of Colorado Cancer Center, Denver, Colorado
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - CCOP - Central Illinois, Decatur, Illinois
  - Veterans Affairs Medical Center - Hines (Hines Junior VA Hospital), Hines, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - CCOP - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Wichita, Wichita, Kansas
  - Veterans Affairs Medical Center - Lexington, Lexington, Kentucky
  - Albert B. Chandler Medical Center, University of Kentucky, Lexington, Kentucky
  - MBCCOP - LSU Medical Center, New Orleans, Louisiana
  - Tulane University School of Medicine, New Orleans, Louisiana
  - Veterans Affairs Medical Center - New Orleans, New Orleans, Louisiana
  - Louisiana State University Health Sciences Center - Shreveport, Shreveport, Louisiana
  - Veterans Affairs Medical Center - Shreveport, Shreveport, Louisiana
  - Boston Medical Center, Boston, Massachusetts
  - Veterans Affairs Medical Center - Boston (Jamaica Plain), Jamaica Plain, Massachusetts
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Veterans Affairs Medical Center - Detroit, Detroit, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - CCOP - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Providence Hospital - Southfield, Southfield, Michigan
  - Veterans Affairs Medical Center - Biloxi, Biloxi, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Veterans Affairs Medical Center - Jackson, Jackson, Mississippi
  - Keesler Medical Center - Keesler AFB, Keesler Air Force Base, Mississippi
  - Veterans Affairs Medical Center - Kansas City, Kansas City, Missouri
  - CCOP - Kansas City, Kansas City, Missouri
  - CCOP - Cancer Research for the Ozarks, Springfield, Missouri
  - St. Louis University Health Sciences Center, St Louis, Missouri
  - CCOP - St. Louis-Cape Girardeau, St Louis, Missouri
  - CCOP - Montana Cancer Consortium, Billings, Montana
  - Veterans Affairs Medical Center - Albuquerque, Albuquerque, New Mexico
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - Herbert Irving Comprehensive Cancer Center, New York, New York
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Veterans Affairs Medical Center - Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic Cancer Center, Cleveland, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Veterans Affairs Medical Center - Dayton, Dayton, Ohio
  - CCOP - Dayton, Kettering, Ohio
  - Oklahoma Medical Research Foundation, Oklahoma City, Oklahoma
  - Veterans Affairs Medical Center - Oklahoma City, Oklahoma City, Oklahoma
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Veterans Affairs Medical Center - Portland, Portland, Oregon
  - CCOP - Columbia River Program, Portland, Oregon
  - CCOP - Greenville, Greenville, South Carolina
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - Simmons Cancer Center - Dallas, Dallas, Texas
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - University of Texas Medical Branch, Galveston, Texas
  - Texas Tech University Health Science Center, Lubbock, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Veterans Affairs Medical Center - San Antonio (Murphy), San Antonio, Texas
  - Veterans Affairs Medical Center - Temple, Temple, Texas
  - CCOP - Scott and White Hospital, Temple, Texas
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Veterans Affairs Medical Center - Salt Lake City, Salt Lake City, Utah
  - CCOP - Virginia Mason Research Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Veterans Affairs Medical Center - Seattle, Seattle, Washington
  - Puget Sound Oncology Consortium, Seattle, Washington
  - CCOP - Northwest, Tacoma, Washington